CLINICAL TRIAL: NCT03370172
Title: A Global, Open-Label, Multicenter, Phase 1/2 Study of the Safety and Dose Escalation of BAX 888, an Adeno-Associated Virus Serotype 8 (AAV8) Vector Expressing B-Domain Deleted Factor VIII (BDD-FVIII) in Severe Hemophilia A Subjects Administered a Single Intravenous Infusion
Brief Title: A Study of BAX 888 in Male Adults With Severe Hemophilia A
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Collaborators: Baxalta Innovations GmbH, now part of Shire (Industry); Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 201501; 2015-005576-22 (EudraCT Number)
Record Dates: First submitted 2017-11-22; First posted 2017-12-12 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: BAX 888 2.0*10^12 cp/kg (Experimental): Cohort 1 participants received a single peripheral intravenous (IV) infusion of BAX 888 at a dose of 2.0*10^12 capsid particles per kilogram (cp/kg) on the day of dosing (Day 0).
  Interventions: Drug: BAX 888
- Cohort 2: BAX 888 6.0*10^12 cp/kg (Experimental): Cohort 2 participants received a single peripheral IV infusion of BAX 888 at a dose of 6.0*10^12 cp/kg on the day of dosing (Day 0).
  Interventions: Drug: BAX 888

INTERVENTIONS:
Drug: BAX 888 — Participants will receive a single peripheral IV infusion of BAX 888 in Cohort 1 and 2 Day 0.
  Other Names: Adeno-associated virus serotype 8 (AAV8) vector expressing B-domain deleted Factor VIII (BDD-FVIII); BAX888

SUMMARY:
The main aim of this study is to check if there are side effects from BAX 888 and to determine the dose of BAX 888 for treating severe hemophilia A in male adults.

Participants will receive one infusion with BAX 888 at the hemophilia treatment center. During the study, participants will visit their study clinic multiple times.

DETAILED DESCRIPTION:
This study consists of 3 cohorts. Participants will be assigned to 1 of 3 dose cohorts with a minimum of 24 hours between dosing of each participant. Initially, 2 participants will be dosed in a cohort, with up to a total of 5 participants if the cohort is expanded based on safety and activity levels data.

Dose escalation: After dosing first 2 participants in cohort 1 the decision will be made on the following: If week 4 FVIII activity levels of both participants are less than (<) 2%, then dose escalation to cohort 2 will be triggered with no further dosing in cohort 1. If FVIII activity levels >=2% are observed in at least 1 participant among the 2 participants the decision to escalate dose or expand the cohort with dosing of additional participants will be based on all available data through Week 14.

Dose expansion: After dose escalation and administration of BAX 888 to the first 2 participants in 3 cohorts: If sustained Week 14 FVIII activity levels are >=30% are not achieved in both participants (first 2 participants in cohorts 1 and 2) then escalation to immediate next cohort will be triggered after Data Monitoring Committee (DMC) review of all available safety and FVIII activity levels data. For cohort 3 dosing of additional participants will be paused until further review of available data. If sustained Week 14 FVIII levels are >=30% in at least 1 of the 2 participants (first 2 participant in cohort 1, 2, 3) then expansion of cohorts 1, 2 (with up to 5 participants), 3 (with up to 3 additional participants) will be initiated with dosing or study could be completed with no further dosing.

23 APRIL 2020: Enrollment of new patients into this study has been paused due to the COVID-19 situation. The duration of this pause is dependent on the leveling and control of the COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 to 75 years at the time of screening.
* Established severe hemophilia A (FVIII:C <1%, measured following >=5 days without FVIII treatment) and/or documented intron 1 inversion or intron 22 inversion mutation in the F8 gene, consistent with severe hemophilia A , and documented evidence of >=3 hemorrhages over the previous 12 months requiring treatment with exogenous FVIII or use of FVIII prophylaxis because of history of frequent bleeding episodes.
* History of greater than (>) 150 exposure days to exogenously administered FVIII concentrates or cryoprecipitate.
* Sexually active men must agree to use barrier contraception (combination of a condom and spermicide) or limit sexual intercourse to post-menopausal, surgically sterilized, or contraception-practicing partners for a minimum of 6 months after administration of BAX 888, or until BAX 888 genomes are no longer detected in the semen, whichever is sooner.
* Participant is willing and able to comply with the requirements of the protocol, including provision of semen samples, maintenance of a diary of bleeding episodes and FVIII protein use.
* Signed informed consent.

Exclusion Criteria:

* Bleeding disorder(s) other than hemophilia A.
* Personal laboratory evidence of having developed inhibitors to FVIII protein at any time (>=0.6 Bethesda units [BU] on any single test).
* Documented prior allergic reaction to any FVIII product.
* Anti-Adeno-associated virus, serotype 8 (AAV8) neutralizing antibody titer >=1:5. Participants whose laboratory assessments are less than or equal to (<=) 1:10 may be re-tested within the same screening window and, if eligibility criterion is met on retest, may be enrolled after confirmation by the Sponsor Medical Monitor.
* Known hypersensitivity to prednisolone or prednisone, or to any of the excipients.
* Having a disease in which treatment with prednisolone or prednisone is not tolerated (including but not limited to osteoporosis with vertebral fractures, difficult to control hypertension, and difficult to control diabetes).
* Evidence of markers of potential underlying risk for autoimmune mediated hepatic disease:

  * Anti-smooth muscle antibody assay results >=40 (Inova QUANTA LiteTM Actin IgG enzyme-linked immunosorbent assay [ELISA]); values of 31 to 39 will be flagged as possibly abnormal and the Investigator and Medical Monitor will evaluate the participant for eligibility.
  * Elevated anti-liver-kidney microsomal antibody type 1 (LKM1) titers.
  * Total immunoglobulin G (IgG) >1.5*upper limit of normal (ULN).
  * Antinuclear antibody (ANA) titer >1:320; OR ANA titer >1:80 if demonstrated concurrently with alanine aminotransferase (ALT) that is >ULN.
* Active Hepatitis virus (Hepatitis C): As indicated by detectable hepatitis C virus (HCV) ribonucleic acid (RNA) by polymerase chain reaction (PCR).
* Hepatitis B: If surface antigen is positive.
* Seropositive for Human Immunodeficiency Virus (HIV).
* Receiving systemic antiviral and/or interferon therapy within 4 weeks prior to enrollment.
* Clinically significant infections (e.g. systemic fungal infections) requiring systemic treatment.
* Known immune disorder (including myeloma and lymphoma).
* Concurrent chemotherapy or biological therapy for treatment of neoplastic disease or other disorders.
* An absolute neutrophil count <1000 cells per cubic millimeter (cells/mm^3).
* Markers of hepatic inflammation or cirrhosis as evidenced by 1 or more of the following:

  * Platelet count of <150,000/microliter (mcL).
  * Serum albumin level is below the central laboratory's lower limit of normal and FibroSURE is >=0.48 (i.e., Metavir staging of F2 or greater). Of note, in participants with a known history of Gilbert's syndrome, a Fibrotest cannot be used for fibrosis testing.
  * Total bilirubin >1.5*ULN and direct bilirubin >=0.5 milligram per deciliter (mg/dL).
  * ALT or aspartate aminotransferase (AST) >1.0*ULN.
  * Alkaline phosphatase (AP) >2.0*ULN.
  * History of liver biopsy indicating moderate or severe fibrosis (Metavir staging of F2 or greater).
  * History of ascites, varices, variceal hemorrhage, or hepatic encephalopathy.
  * Any findings on screening ultrasound that would preclude the safe use of AAV gene therapy.
* Prothrombin time (PT) international normalized ratio (INR) >=1.4.
* Serum creatinine >1.5 mg/dL.
* Urine protein >30 mg/dL or >0.5 gram per day (g/day).
* Body mass index >38.
* Major surgery or an orthopedic surgical procedure planned within 6 months after enrollment.
* Acute or chronic disease that, in the opinion of the investigator, would adversely affect participant safety or compliance or interpretation of study results.
* Received an AAV vector previously or any other gene transfer agent in the previous 12 months prior to Study Day 0.
* Received an investigational intervention or participated in another clinical trial within 4 weeks prior to enrollment or within 5 half-lives of the investigational drug administration, whichever is longer.
* Significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, congestive heart failure, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease).
* Recent history of psychiatric illness or cognitive dysfunction (including drug or alcohol abuse) that in the opinion of the investigator, is likely to impair participants ability to comply with protocol mandated procedures.
* Participant is a family member or employee of the investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2024-07-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (26):
- United States (8):
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Orthopaedic Hospital DBA Orthopaedic Hemophilia Treatment Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - Mount Sinai Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Gulf States Hemophilia and Thrombophilia Center, Houston, Texas
- AKH - Medizinische Universität Wien, Vienna, Austria
- France (8):
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Hôpital Morvan, Brest, Finistere
  - CHU Rennes - Hopital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Tours - Hôpital Trousseau, Tours, Indre Et Loire
  - CHU de Nantes Site Hotel Dieu, Nantes, Loire Atlantique
  - Hopital Jeanne de Flandre - CHU Lille, Lille, Nord
  - Groupement Hospitalier Est- Hôpital Louis Pradel, Bron, Rhone
  - Hôpital Bicêtre, Le Kremlin-Bicêtre, Val De Marne
- Germany (3):
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Vivantes Klinikum im Friedrichshain, Berlin
- Semmelweis Egyetem, Budapest, Hungary
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitari i Politecnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No
Takeda does not provide access to Individual Participant Data when a study is in a very limited (small) study population due to participant privacy concerns such as potential reidentification of study participants.

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fc54db2bf003ab45cf2

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4 participants took part in the study globally from 27 February 2018 to 09 July 2024.
Pre-assignment Details: Participants with severe Hemophilia A participated in the study to receive BAX 888.
Period: Overall Study
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Started | 2 | 2
Completed | 2 | 1
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Safety Set consisted of all participants who received any amount of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (13.44) | 27.5 (3.54) | 28.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With BAX 888-Related Adverse Events (AEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered an investigational product (IP) that does not necessarily have a causal relationship with the treatment. A Serious adverse event (SAE) is an AE resulting in any of the following outcomes: death; life-threatening event; required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. AEs include both serious and non-serious adverse events including development of FVIII inhibitory antibodies, clinically significant changes in standard laboratory parameters, physical exam, and vital signs.
Time Frame: From first dose up to end of the study (approximately 6 years)
Population: The Safety Set consisted of all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
Participants | 2 | 2

2. Secondary Outcome: Change From Baseline in Circulating Plasma FVIII Activity Level
Description: Change from baseline in circulating plasma FVIII activity level, based on one-stage clotting assay was assessed.
Time Frame: Baseline, up to Month 60
Population: The Safety Set consisted of all participants who received any amount of investigational product. Overall number analyzed is the number of participants with data available for analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: International Units per deciliter(IU/dL)
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 1
International Units per deciliter(IU/dL) | 11.40 (1.131) | 248.30 (NA) — Standard Deviation (SD) is not estimable when there is only a single participant.

3. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Circulating Plasma FVIII Antigen Level
Description: Change from baseline in circulating plasma FVIII antigen (protein) levels were to be assessed and number of participants with clinically significant change as determined by the principal investigator (PI) were reported.
Time Frame: Baseline, up to Month 60
Population: The Safety Set consisted of all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
Participants | 2 | 0

4. Secondary Outcome: Annualized Bleed Rate (ABR)
Description: ABR in comparison to before gene transfer will be assessed. A bleed is defined as subjective or objective evidence of bleeding which may or may not require treatment with FVIII. ABR was calculated as (number of bleeding episodes/observed treatment period in days)*365.25.
Time Frame: Up to approximately 6 years 4 months
Population: The Safety Set consisted of all participants who received any amount of investigational product.
Measure: Mean (Standard Deviation); unit: bleeds per year
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
bleeds per year | 1.0 (1.41) | 0.5 (0.71)

5. Secondary Outcome: Percentage of Participants With a Reduction in Consumption of Exogenous FVIII
Description: The reduction in consumption of exogenous FVIII was assessed by comparing the amount of exogenous FVIII taken at earliest time point available (prior to BAX 888 infusion) with the amount taken at the last post-infusion timepoint available, during the study. Percentage of participants with reduction in consumption of exogenous FVIII are reported.
Time Frame: Up to approximately 6 years 4 months
Population: The Safety Set consisted of all participants who received any amount of investigational product.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
percentage of participants | 0.0 | 0.0

6. Secondary Outcome: Number of Participants Who Developed Inhibitory Antibodies to FVIII
Description: Participants were assessed to check if they developed inhibitory antibodies to FVIII.
Time Frame: Up to approximately 6 years 4 months
Population: The Safety Set consisted of all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

7. Secondary Outcome: Number of Participants Who Developed Total Binding Antibodies to FVIII
Description: Participants were assessed to check if they developed total binding antibodies to FVIII (Immunoglobulin G [IgG], Immunoglobulin M [IgM]).
Time Frame: Up to approximately 6 years 4 months
Population: The Safety Set consisted of all participants who received any amount of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Humoral and Cell-Mediated Immune Response to AAV8 and FVIII Proteins
Description: The humoral (antibody-mediated) and cell-mediated immune response to adeno-associated virus (AAV8) (the vector) and FVIII proteins, was assessed. Humoral Immune Response: It is indicated by presence of specific antibodies. The anti-AAV8 binding antibodies, IgG or IgM were measured by the enzyme-linked immunosorbent assay (ELISA) method. Neutralizing antibodies were measured by a cell-based luminescent assay. Cell-mediated Immune response: The AAV8 and FVIII specific cell mediated immunity was assessed using validated interferon-γ (IFN-γ) enzyme-linked immunosorbent spot (ELISpot) assays. This assay tests the human T-cell recall response to the AAV8 and FVIII proteins. These proteins were called antigens for these tests (AAV8 peptide pools 1, 2, 3 and two pooled test antigens (1 and 2) for FVIII). Number of participants who had humoral and/or cell mediated immune response to AAV8 and FVIII proteins, are reported by humoral and cell mediated immune response categories.
Time Frame: Up to approximately 6 years 4 months
Population: The Safety Set consisted of all participants who received any amount of investigational product. Number analyzed is the number of participants with data available for analysis for the specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
Participants
  Humoral: Binding Ab to AAV8 IgG Titer: number analyzed (Participants) | 2 | 1
  Humoral: Binding Ab to AAV8 IgG Titer | 2 | 1
  Humoral: Binding Ab to AAV8 IgM Titer: number analyzed (Participants) | 0 | 0
  Humoral: Neutralising Ab to AAV8 Titer: number analyzed (Participants) | 2 | 1
  Humoral: Neutralising Ab to AAV8 Titer | 2 | 1
  Cell-Mediated: AAV8 Peptide Pool 1 Mean: number analyzed (Participants) | 2 | 1
  Cell-Mediated: AAV8 Peptide Pool 1 Mean | 0 | 1
  Cell-Mediated: AAV8 Peptide Pool 2 Mean: number analyzed (Participants) | 2 | 1
  Cell-Mediated: AAV8 Peptide Pool 2 Mean | 1 | 1
  Cell-Mediated: AAV8 Peptide Pool 3 Mean: number analyzed (Participants) | 2 | 1
  Cell-Mediated: AAV8 Peptide Pool 3 Mean | 1 | 1
  Cell-Mediated: FVIII Peptide Pool 1 Mean: number analyzed (Participants) | 2 | 1
  Cell-Mediated: FVIII Peptide Pool 1 Mean | 0 | 0
  Cell-Mediated: FVIII Peptide Pool 2 Mean: number analyzed (Participants) | 2 | 1
  Cell-Mediated: FVIII Peptide Pool 2 Mean | 1 | 1

9. Secondary Outcome: Surveillance of AAV8 Genome Shedding
Description: Surveillance of AAV8 genome shedding in blood, saliva, semen, stool and urine until two consecutive negative results were assessed.
Time Frame: Blood: Day 1, weekly at Clinic Visits between Weeks 1-15, and at Months 4 and 5; Saliva, Semen, and Stool: Day 1 and Week 1; Urine: Day 1 and Weeks 1,2,3
Population: The Safety Set consisted of all participants who received any amount of investigational product. The data was collected for each category until 2 consecutive measurements were negative. Number analyzed is the number of participants with data available for analysis at specified time points.
Measure: Mean (Standard Deviation); unit: Genome copies per 100 ng of sample
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
Number analyzed (Participants) | 2 | 2
Genome copies per 100 ng of sample
  Blood: Day 1: number analyzed (Participants) | 0 | 1
  Blood: Day 1 |  | 3684434.0 (NA) — SD was not estimable for a single participant.
  Blood: Week 1: number analyzed (Participants) | 1 | 2
  Blood: Week 1 | 3634.0 (NA) — SD was not estimable for a single participant. | 18608.0 (664.68)
  Blood: Week 2 | 2076.0 (295.57) | 10670.0 (3900.40)
  Blood: Week 3 | 2069.0 (741.05) | 9845.0 (6488.41)
  Blood: Week 4: number analyzed (Participants) | 1 | 2
  Blood: Week 4 | 1098.0 (NA) — SD was not estimable for a single participant. | 9033.5 (4978.74)
  Blood: Week 5 | 1483.0 (1097.43) | 7884.0 (288.50)
  Blood: Week 6 | 904.0 (335.17) | 5372.5 (441.94)
  Blood: Week 7 | 1004.0 (656.20) | 6808.0 (1121.47)
  Blood: Week 8 | 828.5 (267.99) | 7384.0 (1011.16)
  Blood: Week 9 | 714.5 (222.74) | 6384.5 (195.87)
  Blood: Week 10 | 773.0 (9.90) | 6144.5 (939.74)
  Blood: Week 11 | 755.0 (241.83) | 3935.0 (1547.15)
  Blood: Week 12 | 728.0 (130.11) | 3893.5 (276.48)
  Blood: Week 13 | 654.0 (22.63) | 3044.5 (1191.47)
  Blood: Week 14 | 735.5 (82.73) | 2856.0 (1473.61)
  Blood: Week 15: number analyzed (Participants) | 1 | 2
  Blood: Week 15 | 742.0 (NA) — SD was not estimable for a single participant. | 2812.0 (2083.14)
  Blood: Month 4: number analyzed (Participants) | 2 | 1
  Blood: Month 4 | 422.0 (192.33) | 3066.0 (NA) — SD was not estimable for a single participant.
  Blood: Month 5: number analyzed (Participants) | 0 | 1
  Blood: Month 5 |  | 210.0 (NA) — SD was not estimable for a single participant.
  Saliva: Day 1 | 935.0 (268.70) | 2076.5 (473.05)
  Saliva: Week 1: number analyzed (Participants) | 0 | 2
  Saliva: Week 1 |  | 352.5 (12.02)
  Semen: Day 1: number analyzed (Participants) | 1 | 2
  Semen: Day 1 | 55.0 (NA) — SD was not estimable for a single participant. | 230.5 (188.80)
  Semen: Week 1: number analyzed (Participants) | 0 | 1
  Semen: Week 1 |  | 194.0 (NA) — SD was not estimable for a single participant.
  Stool: Day 1: number analyzed (Participants) | 0 | 1
  Stool: Day 1 |  | 5985.0 (NA) — SD was not estimable for a single participant.
  Stool: Week 1: number analyzed (Participants) | 0 | 2
  Stool: Week 1 |  | 7164.0 (7993.14)
  Urine: Day 1 | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection. | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection.
  Urine: Week 1 | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection. | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection.
  Urine: Week 2 | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection. | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection.
  Urine: Week 3 | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection. | NA (NA) — Mean and SD were not estimable due to genome concentrations being Below Limit of Detection.

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to approximately 6 years 4 months; SAEs and Other (Non-Serious) AEs: From first dose up to end of the study (approximately 6 years)
Description: The Safety Set consisted of all participants who received any amount of investigational product.
Arm/Group | Cohort 1: BAX 888 2.0*10^12 cp/kg | Cohort 2: BAX 888 6.0*10^12 cp/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BAX 888 2.0*10^12 cp/kg (N=2) | Cohort 2: BAX 888 6.0*10^12 cp/kg (N=2)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: BAX 888 2.0*10^12 cp/kg (N=2) | Cohort 2: BAX 888 6.0*10^12 cp/kg (N=2)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Headache (Nervous system disorders) | 1 | 1
Hyperphagia (Metabolism and nutrition disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Initial insomnia (Psychiatric disorders) | 0 | 1
Irritability (Psychiatric disorders) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
SARS-CoV-2 test positive (Investigations) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Tongue geographic (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Weight increased (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-11-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT03370172/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT03370172/SAP_001.pdf